CLINICAL TRIAL: NCT02973555
Title: Can Platelet-rich Plasma (PRP) Promote Endometrial Growth and Improve Pregnancy Outcome of Patients With Thin Endometrium Undergoing Assisted Reproductive Technology (ART) Treatments?
Brief Title: Platelet-Rich Protein and the Endometrium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP-HMO-CTIL
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRP injection (Experimental)
  Interventions: Other: PRP injection

INTERVENTIONS:
Other: PRP injection — autologous intrauterine infusion of PRP

SUMMARY:
Platelet-rich plasma (PRP) may promote the endometrial growth and improve pregnancy outcome of patients with thin endometrium undergoing ART treatments.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a frozen thawed embryo transfer cycle with poor endometrial response to estrogen (< 7 mm) after at least two standard preparation protocols, of which one was canceled due to thin endometrium

Exclusion Criteria:

* none

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
endometrial thickness >7mm | 1 month

SECONDARY OUTCOMES:
Positive serum pregnancy test | 14 days post embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Kochman, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No